CLINICAL TRIAL: NCT03719989
Title: A Phase II Study of Epigenetic Priming Using Azacitidine Followed by Rituximab-GDP Immunochemotherapy in Patients With Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Brief Title: Azacitidine and Rituximab-GDP Immunochemotherapy in Patients With Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Acronym: EPIC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sung-Soo Yoon, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPIC
Record Dates: First submitted 2018-10-15; First posted 2018-10-25 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Diffuse Large B Cell Lymphoma; Relapsed Non Hodgkin Lymphoma; Refractory Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): This study is sing-arm study. Therefore, all enrolled patients will be treated with azacitidine plus R-GDP regimen
  Interventions: Drug: azacitidine plus R-GDP

INTERVENTIONS:
Drug: azacitidine plus R-GDP — azacitidine S.C 25 mg/m2 D1,2,3,4,5 rituximab I.V. 375 mg/m2 D8 gemcitabine I.V. 1,000 mg/m2, D8,15 dexamethasone I.V. or P.O. 40 mg D8,9,10,11 every 21 days, up to 6 cycles
  Other Names: N/E

SUMMARY:
This phase II clinical trial aims at evaluating the efficacy and safety of azacitidine followed by rituximab-GDP immunochemotherapy in patients with relapsed/refractory diffuse large B-cell lymphoma (DLBCL). Patients who were treated with from 1 to 4 lines of prior therapies for relapsed/refractory DLBCL wee eligible. azacitidine will be treated one week prior to conventional rituximab-gemcitabine, dexamethasone, cisplatin (R-GDP) immunochemotherapy. Patients will be treated every 21 days as one cycle, and up to 6 cycles. The primary endpoint of this study is objective response rate according to the Lugano response criteria for non-Hodgkin lymphoma, and secondary endpoints are safety, complete response, progression-free survival, and overall survival.

DETAILED DESCRIPTION:
This phase II clinical trial aims at evaluating the efficacy and safety of azacitidine followed by rituximab-GDP immunochemotherapy in patients with relapsed/refractory diffuse large B-cell lymphoma (DLBCL). This study is designed with the expectation of correction of aberrant hypermethylation of tumor suppressor genes by preceding use of low dose azacitidine thereby re-sensitizing chemosensitivity of tumor cells. Patients who were treated with from 1 to 4 lines of prior therapies for relapsed/refractory DLBCL wee eligible. Planned initial doses of the current regimen are as follows;

azacitidine S.C 25 mg/m2 D1,2,3,4,5 rituximab I.V. 375 mg/m2 D8 gemcitabine I.V. 1,000 mg/m2, D8,15 dexamethasone I.V. or P.O. 40 mg D8,9,10,11 cisplatin 70 mg/m2 I.V. D8

Patients will be treated every 21 days as one cycle, and up to 6 cycles of treatment will be conducted. Especially, first 3~6 patients will be regarded as 'lead-in safety cohort' and their safety will be reviewed by an independent data and safety monitoring board (DSMB). The primary endpoint of this study is objective response rate according to the Lugano response criteria for non-Hodgkin lymphoma, and secondary endpoints are safety, complete response, progression-free survival, and overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. age from 19 to 75 years
2. diagnosed as diffuse large B-cell lymphoma according to the World Health Organization 2016 criteria
3. with any measurable lesion by radiologic studies (direct measurement is allowed in cases of (sub)cutaneous lesions)
4. patients who were initially treated with rituximab plus cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) or other rituximab-containing immunochemotherapy and relapsed or refractory to prior treatment
5. previously treated with from1 to 4 lines of therapy

   * autologous stem cell transplant (ASCT) will be counted as 1 line of therapy
   * in cases of previously treated with ASCT, patients 1) who elapsed at 60 days and 2) who have lower risk of severe bone marrow suppression and infectious complication, judged by physician
6. ASCT ineligible or no further plan of ASCT due to previous transplantation
7. Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0~2
8. Hb ≥ 8.0 g/dL, absolute neutrophil count (ANC) ≥ 1,000/mm3, Platelet ≥ 100,000/mm3 prior to enrollment

   * correction of Hb by transfusion will be allowed
   * in cases of bone marrow involvement, patients will be included if they have ANC ≥ 500/mm3, Platelet ≥ 50,000/mm3 and no significant infection risk or transfusion dependency
9. Glomerular Filtration Rate > 60 mL/min calculated according to Cockcroft-Gault or Modification of Diet in Renal Disease (MDRD) equation, and total bilirubin < 2.5 mg/dL, aspartate amino-transferase (AST) and alanine amino- transferase (ALT) < x3 upper limit of normal (ULN)

   * In cases of hepatic involvement of DLBCL, AST or ALT < x5 ULN will be allowed
   * In cases of Gilbert syndrome, Direct bilirubin < 2.5 ULN will be allowed
10. patients who agree to do highly effective contraception during and 3 months after treatment
11. patients who agree not to be pregnant or breast-feeding and had a negative result for screening pregnancy test
12. life expectancy > 3 months

Exclusion Criteria:

1. primary or secondary central nervous system DLBCL
2. patients with or strongly suggestive of lymphomatous involvement on eye, epidural area, kidney/adrenal gland, breast, testes, or uterus
3. intravascular DLBCL
4. DLBCL transformed from low grade lymphoma
5. high grade B-cell lymphomas other than DLBCL: primary mediastinal large B-cell lymphoma, high-grade B-cell lymphoma not otherwise specified (NOS), high-grade B-cell lymphoma with myelocytomatosis oncogene (MYC) and/or B-cell lymphoma 6 (BCL6) rearrangements, B-cell lymphoma, unclassifiable with features intermediate between DLBCL and classical Hodgkin lymphoma
6. human immunodeficiency virus (HIV) associated DLBCL
7. patients with liver cirrhosis of Child-Pugh Classification B or higher, or active hepatitis B (HBV) or hepatitis C (HCV) infection

   * in cases of patients who are positive for HBsAg or HBcAb immunoglobulin G (IgG) but no evidence of active infection, patients who are negative for HBV DNA will be allowed only with adequate anti-viral prophylaxis
   * in cases of patients who are positive for hepatitis C antibody, patients will be allowed if they satisfy all other inclusion criteria and without evidence of liver cirrhosis (irrespective of HCV RNA titer)
   * patients who were diagnosed HCV less than 6 months before screening period will be excluded unless they have negative result for HCV RNA
8. patients with active infection treated with anti-microbial agents
9. patients who were diagnosed malignancy other than lymphoma, either actively treated or have been received chemotherapy or radiation therapy less than 3 years from the time of enrollment
10. Major surgery within 21 days (open laparotomy for diagnostic biopsy will be exempted)
11. patients who underwent hypersensitivity, severe allergic reaction or anaphylaxis to rituximab or other chimeric/humanized antibodies
12. patients who underwent hypersensitivity, severe allergic reaction or anaphylaxis gemcitabine, azacitidine, or cisplatin
13. severe congestive heart failure, unstable heart or pulmonary diseases
14. pregnant or lactating women
15. during radiation therapy to chest area (considering previous reports of severe esophagitis and pneumonitis after concurrent chemoradiation with gemcitabine)
16. with any prior experience of posterior reversible encephalopathy syndrome or progressive multifocal leukoencephalopathy due to rituximab
17. with any prior experience of Stevens-Jones syndrome or toxic epidermal necrosis

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | up to 3 years
  according to Lugano response criteria for non-Hodgkin lymphoma

SECONDARY OUTCOMES:
Safety (adverse events and severe adverse events) | up to 3 years
  according to CTCAE V4.03 criteria
Complete response rate | up to 3 years
  according to Lugano response criteria for non-Hodgkin lymphoma
Progression-free survival | up to 3 years
  From date of enrollment until date of first documented progression or date of death from any cause, whichever came first
Overall survival | up to 3 years
  From date of enrollment until date of death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim DH, Kong JH, Hong J, Byun JM, Shin DY, Koh Y, Kim I, Park J, Do YR, Kim JA, Kim WS, Shin HJ, Yoon SS. Azacitidine followed by R-GDP in transplant-ineligible relapsed/refractory diffuse large B-cell lymphoma: preliminary results from a multicenter, phase II study. Ther Adv Hematol. 2025 Jul 11;16:20406207251349361. doi: 10.1177/20406207251349361. eCollection 2025. PMID 40656663